CLINICAL TRIAL: NCT00954577
Title: The Pathogenesis of Type 2 Diabetes in Children and Utility of a School-based Intervention to Reduce Obesity and Diabetes in Children
Brief Title: Reduce Obesity and Diabetes
Acronym: ROAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academy for Medical Development and Collaboration, New York (Other)
Responsible Party: Maria Mitchell, Ph.D., President, AMDeC
Other Study IDs: amdecroad
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabetes; Pediatric Obesity; Dyslipidemia
Keywords: obesity; diabetes; exercise; education; child
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Pediatric Obesity; Dyslipidemias; Obesity; Diabetes Mellitus; Motor Activity | interventions — Nutritional Status; Health

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Nutrition, health, and exercise education — The classroom intervention is part of the routine science curriculum and consists of 14 sessions taught by the investigators. Topics covered include the development of type 2 diabetes, nutrition education, exercise education, and overall healthy lifestyle education (both at home and in school). The intervention is offered in each year to all grades and to all students, regardless of whether or not they are enrolled in the study. The exercise intervention is optional and consists of 2-3 sessions per week of aerobic exercise (dancing) taught by pediatric trainers and offered in lieu of regular gym classes.

SUMMARY:
This study examines risk factors for type 2 diabetes in children representing multiple discrete ethnic groups. It also examines the short term effects of school-based health education supervised exercise on metabolic risk factors for type 2 diabetes mellitus in children. The investigators hypothesize that exercise and health education will significantly improve insulin sensitivity in all children, especially in children who are already insulin resistant, thereby lowering the risk that they will go on to develop type 2 diabetes mellitus. The specific hypotheses being tested are:

1. Insulin resistance will be most evident in overweight children while an impaired ability of the pancreas to release insulin will be most evident in children with a family history of type 2 diabetes mellitus.
2. Exercise will significantly improve insulin resistance (as measured by the fasting glucose/insulin ratio) with little effect on insulin secretory capacity in children.
3. Participation in a school-based health, nutrition, and exercise education program will have long term beneficial effects on health related behaviors and on insulin resistance in all children, regardless of their level of diabetes risk.

DETAILED DESCRIPTION:
The prevalence of type 2 diabetes mellitus (type 2 DM) among adolescents has increased > 10 fold over the past decade. Type 2 DM reflects the interactions of genes/traits conveying an increased risk of impaired function of the pancreatic cells that secrete insulin (islet cells)and muscle/liver insulin sensitivity with environmental factors such as reduced levels of activity and increasing adiposity. Both impaired islet cell function and insulin resistance are independently associated with increased risk of subsequent diabetes mellitus and may be considered as 'prediabetic' phenotypes. This study examines the prevalence of prediabetic phenotypes and the effects of supervised exercise/nutrition education on risk factors for type 2 DM in 6th-8th grade students who will undergo a 5 minute intravenous glucose tolerance test, as well as measurements of other diabetes risk factors including family history, body composition, circulating concentrations of molecules (cytokines) that are markers of inflammation , and lipid profiles, before and after participating in the intervention. These studies will also be used to calculate both the ability of the pancreas to secrete insulin and the sensitivity of the students to insulin. No previous studies have isolated the effects of exercise and nutrition education on different diabetes subphenotypes in children. To insure the necessary ethnic diversity necessary to these studies, data will be pooled in a multisite study with Mt. Sinai, North Shore/LIJ, Maimonides, and Winthrop Hospitals. We will remain in contact with students to track subsequent development of diabetes intervention effects on lifestyle. We hypothesize that diabetes risk in most students will be reduced by exercise and education in a healthy lifestyle but that the type of health benefit (i.e., improved body fatness, improved insulin sensitivity, improved insulin secretion, improved cholesterol, or decreased inflammation) will be different between ethnic groups. The results of these studies will, we believe, demonstrate the benefits of health and physical education programs to all students, regardless of diabetes risk, and will also enable us to better understand how diabetes develops in children and what expectations we can have for health improvement in different ethnic groups from such an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children in 6th-8th grade

Exclusion Criteria:

* Diabetes
* Exercise induced asthma
* Pregnancy
* Any chronic medication that interferes with glucose homeostasis

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children in 6th-8th grade.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-07; Primary Completion 2012-05 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in diabetes risk factors including insulin secretory capacity, insulin sensitivity, body fat content, dyslipidemia, and circulating concentrations of pro-inflammatory cytokines. | In December and May of each school year

SECONDARY OUTCOMES:
Improvement in self-esteem and in health-related behaviors. | December and May of each school year

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Maimonides Medical Center, Brooklyn, New York
  - North Shore LIJ Schneider Children's Hospital, Manhasset, New York
  - Winthrop University Hospital, Mineola, New York
  - Mt. Sinai Medical Center, New York, New York
  - Columbia University Medical Center/The New York Presbyterian Hospital, New York, New York

REFERENCES:
- [Background] Rosenbaum M, Nonas C, Horlick M, Fennoy I, Vargas I, Schachner H, Kringas P, Stanton K, Weil R; Camino Diabetes Prevention Group. beta-Cell function and insulin sensitivity in early adolescence: association with body fatness and family history of type 2 diabetes mellitus. J Clin Endocrinol Metab. 2004 Nov;89(11):5469-76. doi: 10.1210/jc.2004-0971. PMID 15531499
- [Result] Rosenbaum M, Nonas C, Weil R, Horlick M, Fennoy I, Vargas I, Kringas P; Camino Diabetes Prevention Group. School-based intervention acutely improves insulin sensitivity and decreases inflammatory markers and body fatness in junior high school students. J Clin Endocrinol Metab. 2007 Feb;92(2):504-8. doi: 10.1210/jc.2006-1516. Epub 2006 Nov 7. PMID 17090635